CLINICAL TRIAL: NCT04872673
Title: The Professional Values and Ethical Sensitivities of Turkish Senior Nursing Students in Distance Education During the COVID-19 Pandemic
Brief Title: The Professional Values and Ethical Sensitivities During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Ayşegül Akca (Other)
Responsible Party: Sponsor-Investigator, Ayşegül Akca, Research Assistant, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Other Study IDs: 42/2020
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Professional Values; Ethical Sensitivities
Keywords: COVID-19; ethical sensitivity; nursing student; professional value
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted to examine the professional values and ethical sensitivities of senior nursing students in distance education during the COVID-19 pandemic. During the COVID-19 process, senior nursing students continue their education with distance education practices. The sample consisted of 302 senior nursing students.

ELIGIBILITY:
Inclusion Criteria:

* being over the age of 18
* being a fourth level student
* agreed to participate in the research

Exclusion Criteria:

* being diagnosed with a neuropsychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: senior nursing students
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
The first evaluation- Pre-test | February-2020
  the Nurses Professional Values Scale-Revised Score (The total score obtained from the scale varies between 26 and 130. A high score indicates strong adherence to professional values.)
The first evaluation- Pre-test | February-2020
  Modified Moral Sensitivity Questionnaire for Student Nurses Score (The total score obtained from the scale is between 30 and 210. A high score indicates high ethical sensitivity.)
The second evaluation- Post-test | July-2020
  the Nurses Professional Values Scale-Revised Score (The total score obtained from the scale varies between 26 and 130. A high score indicates strong adherence to professional values.)
The second evaluation- Post-test | July-2020
  Modified Moral Sensitivity Questionnaire for Student Nurses Score (The total score obtained from the scale is between 30 and 210. A high score indicates high ethical sensitivity.)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)